CLINICAL TRIAL: NCT04467853
Title: A Phase 1, Open-Label Study Evaluating the Safety, Tolerability and Efficacy of LCAR-C18S, an CAR-T Cell Therapy Targeting Claudin18.2 in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study to Evaluate CAR-T Cell-based Medicinal Product in the Treatment of Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Both the sponsors and collaborator are considering terminating the study
Sponsor: Shanghai East Hospital (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Principal Investigator, Jin Li, Director, Shanghai East Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM2L201910
Record Dates: First submitted 2020-07-01; First posted 2020-07-13 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-C18S Cells (Experimental): Each subject will receive LCAR-C18S Cells
  Interventions: Biological: LCAR-C18S cells

INTERVENTIONS:
Biological: LCAR-C18S cells — Before treatment with LCAR-C18S cells, subjects will receive a conditioning regimen

SUMMARY:
This is a prospective, single-arm, open-label Phase 1 dose-finding and expansion study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy profiles of the cell-based LCAR-C18S (hereinafter "LCAR-C18S") in subjects with Claudin18.2-positive advanced solid Tumors.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label Phase 1 dose-finding and expansion study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor efficacy profiles of the cell-based LCAR-C18S (hereinafter "LCAR-C18S") in subjects with Claudin18.2-positive advanced solid Tumors. Patients who meet the eligibility criteria will receive LCAR-C18S infusion. The study will include the following sequential phases: screening, pre-treatment , treatment and follow up

ELIGIBILITY:
Inclusion Criteria:

1. The subjects have been fully informed of the possible risks and benefits of participating in the study and have signed the informed consent form;
2. Age 18-70 years;
3. Immunohistochemistry of tumor tissue samples indicates Claudin18.2 positive ;
4. Recurrent or metastatic advanced solid tumors (including advanced gastric cancers and non-gastric cancers) and have been failed to prior lines of systemic treatment
5. According to the RECIST v1.1, at least one measuable tumor lesion;
6. ECOG performance status score of 0-1;
7. Expected survival ≥ 3 months;
8. Subjects should have adequate organ functions before screening and treatment.
9. Women of childbearing age must have a negative blood pregnancy test; subjects of childbearing potential must use effective contraception for ≥ 1 year after the final study treatment.

Exclusion Criteria:

1. Previous CAR-T cell therapy or other cell therapies or therapeutic tumor vaccination against any target;
2. Any previous therapy targeting Claudin18.2;
3. Prior antitumor therapy with insufficient washout period;
4. Pregnant or lactating women;
5. Brain metastases with central nervous system symptoms;
6. Uncontrolled diabetes;
7. Oxygen is required to maintain adequate blood oxygen saturation;
8. Gastric perforation, pyloric obstruction, complete biliary obstruction, complete or incomplete intestinal obstruction requiring clinical intervention, or pleural effusion or peritoneal effusion requiring clinical intervention;
9. Clinically significant liver disorders (including liver cirrhosis, active viral hepatitis or other hepatitis);
10. HIV, Treponema pallidum or HCV serologically positive;
11. Severe underlying disease
12. New York Heart Association (NYHA) Class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50%; unstable angina, myocardial infarction or coronary artery bypass grafting (CABG) in the past 6 months; history of severe non-ischemic cardiomyopathy; or severe uncontrolled arrhythmia;
13. Any condition that, in the opinion of the investigator, will make the subject unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and incidence, severity, and type of treatment-emergent adverse events (TEAEs),Safety | Minimum 2 years after LCAR-C18S infusion (Day 1)
  Dose-limiting toxicity (DLT) and incidence, severity, and type of treatment-emergent adverse events (TEAEs),Safety
To determine the recommended dose of the phase Ⅱ trial of this cell therapy (RP2D) | 90 days post infusion
  To determine the recommended dose of the phase Ⅱ trial of this cell therapy (RP2D)
Pharmacokinetic (PK) parameters | Minimum 2 years after LCAR-C18S infusion (Day 1)
  Blood samples will be collected for determination of cellular concentrations and transgenic levels of serum LCAR-C18S for pharmacokinetic analysis

SECONDARY OUTCOMES:
Overall response rate (ORR) after administration | Minimum 2 years after LCAR-C18S infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LCAR-C18S cell infusion, and the objective tumor response rate will be calculated for patients with measurable disease per RECIST 1.1 only
Progress Free Survival (PFS) after administration | Minimum 2 years after LCAR-C18S infusion (Day 1)
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LCAR-C18S to the first documented disease progression (according to RECIST 1.1) or death (due to any cause), whichever occurs first
Overall Survival (OS) after administration | Minimum 2 years after LCAR-C18S infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LCAR-C18S to death of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, PhD, Principal Investigator — Shanghai East Hospital
Locations (3):
- China (3):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Shanghai East Hospital, Shanghai, China/Shanghai
  - Shanghai Artemed Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No